CLINICAL TRIAL: NCT04896268
Title: Prospective, Multicentric, Randomized, Open-label Study Comparing the Efficacy, in Terms of Quality of Life, and Safety of RAdiofrequency Versus HAL- RAR DOppler in Hemorrhoidal Pathology
Brief Title: Efficacy and Safety of RAdiofrequency Versus HAL- RAR DOppler in Hemorrhoidal Pathology
Acronym: RADO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RADO study
Record Dates: First submitted 2021-05-17; First posted 2021-05-21 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Echocardiography, Doppler

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, therapeutic, comparative, parallel group, randomised controlled open-label, superiority, single-centre, national study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency (Experimental): Rafaelo's technique consists of delivering a low temperature 4 MHz radiofrequency wave current into the haemorrhoidal vascular tissue using a large single-use needle with microfibre electrodes at the end. The intracellular water in the tissue and the injection of a locally injectable Xylocaine cushion serve as resistance to the vaporisation waves without releasing water vapour, thus avoiding the damage usually encountered in electrosurgery. The delayed phenomenon is cell volatilisation. Vaporisation of the tissue allows significant haemostasis without burns. Tissue changes will depend directly on the temperature emitted and the duration of exposure to the radiofrequence current. The fibrosis process starts during the session and continues for several days to weeks, allowing the reduction of the haemorrhoidal cushions.
  Interventions: Device: Radiofrequency
- Arterial ligation then recto-anal repair with Doppler (Active Comparator): Arterial ligation aims to "de-arterialise" the haemorrhoids by selectively decreasing the arterial flow of the haemorrhoidal plexuses while avoiding obstructing the venous return. It is distinguished from mucopexy or recto anal repair (RAR®) which fixes the prolapsed hemorrhoidal plexus. Instead of excising the haemorrhoids, the principle is to reduce their size and to restore the anatomical relationships of the haemorrhoidal plexuses in the anal canal.
  Interventions: Device: Arterial ligation then recto-anal repair with Doppler

INTERVENTIONS:
Device: Radiofrequency — Rafaelo's technique consists of delivering a low-temperature 4 MHz radiofrequency wave current into the haemorrhoidal vascular tissue using a large single-use needle with microfibre electrodes at the end.
  Arms: Radiofrequency
Device: Arterial ligation then recto-anal repair with Doppler — The aim of arterial ligation is to "de-arterialise" the haemorrhoids by reducing the arterial flow of the haemorrhoidal plexuses while avoiding obstructing the venous return.
  Arms: Arterial ligation then recto-anal repair with Doppler

SUMMARY:
Haemorrhoids are composed of tissue rich in blood vessels and are present in all individuals inside the anus (internal haemorrhoids) or under the skin of the anus (external haemorrhoids). Haemorrhoidal disease (HD) occurs when haemorrhoids become troublesome and cause symptoms such as pain, bleeding, prolapse or oozing. In case of failure of medical treatment, instrumental procedures or extensive disease, surgical treatment can be considered. There are two classic surgical techniques. The first is the pedicle haemorrhoidectomy of the Milligan and Morgan type. The second classic surgical technique is the Longo stapled anopexy. Recently, less invasive surgical techniques such as arterial ligation (HAL, with or without Doppler) followed by recto-anal repair (RAR for "Recto Anal Repair") and sometimes associated with mucopexy, which allows the excess mucosa to be ligated and the muco-haemorrhoidal tissue to be fixed to the rectal wall, have developed. The use of radiofrequency current (Rafaelo technique) in the treatment of haemorrhoidal disease is an innovative technique of haemorrhoidal thermocoagulation. It is a mini-invasive technique, which can be performed under sedation or short general anaesthesia (GA), with little pain, allowing a rapid return to normal life and a short time off work. Although this technique is already used in other European countries: Poland, Germany, Belgium, Great Britain (UK), there is now a Polish, German, Spanish and English study in the process of publication. There have been no studies in France to evaluate this new technique and assess its good tolerance, the duration of work stoppage, the improvement in quality of life and the evaluation of its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female consulting for hemorrhoidal pathology (grade II or III) after failure of medico-instrumental treatments.
* Age ≥ 18 years and < 75 years
* Mandatory affiliation to a health insurance system.
* Patient having been informed of the study and having given informed consent

Exclusion Criteria:

* Patients with chronic inflammatory bowel disease
* Patients with suspected gastro-colic pathology
* Haematological diseases
* Anal fistulas
* Patients unable to discontinue anti-vitamin K or oral anticoagulants
* Associated anal fissure
* External haemorrhoidal disease
* Pregnant or breastfeeding women
* Patients under legal protection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
To demonstrate an increase in quality of life, at 1 month post-procedure, when haemorrhoidal disease is managed with radiofrequency versus HAL-RAR with Doppler | 1-month visit
  The Haemorrhoidal Disease and Anal Fissure questionnaire

SECONDARY OUTCOMES:
Pain evaluation | 1-month visit
  Numerical scale (minimum: 0; maximum: 10)
Pain evaluation | 6-month visit
  Numerical scale (minimum: 0; maximum: 10)
feasibility of the 2 techniques under simple antiplatelet agents, anti-vitamin K or oral anticoagulant. | 6-month visit
  Success rate of radiofrequency procedure to be compared between patients taking or not taking AAP, AOD or VKA
Occurrence of a relapse | through study completion, an average of 6 months
  date of relapse, if relapse
Recording of specific symptoms that indicate improvement in hemorrhoidal disease | through study completion, an average of 6 months
  Occurrence of bleeding / prolapse
Time to return to work | through study completion, an average of 6 months
  Duration of work interruption (in days)
Safety evaluation | through study completion, an average of 6 months
  Adverse event

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Private hospital Guillaume de Varye, Saint-Doulchard
  - Centre Clinical, Soyaux

REFERENCES:
- [Background] Aigner F, Bodner G, Gruber H, Conrad F, Fritsch H, Margreiter R, Bonatti H. The vascular nature of hemorrhoids. J Gastrointest Surg. 2006 Jul-Aug;10(7):1044-50. doi: 10.1016/j.gassur.2005.12.004. PMID 16843876
- [Background] Brown SR, Tiernan JP, Watson AJM, Biggs K, Shephard N, Wailoo AJ, Bradburn M, Alshreef A, Hind D; HubBLe Study team. Haemorrhoidal artery ligation versus rubber band ligation for the management of symptomatic second-degree and third-degree haemorrhoids (HubBLe): a multicentre, open-label, randomised controlled trial. Lancet. 2016 Jul 23;388(10042):356-364. doi: 10.1016/S0140-6736(16)30584-0. Epub 2016 May 25. PMID 27236344
- [Background] Loder PB, Kamm MA, Nicholls RJ, Phillips RK. Haemorrhoids: pathology, pathophysiology and aetiology. Br J Surg. 1994 Jul;81(7):946-54. doi: 10.1002/bjs.1800810707. PMID 7922085
- [Background] Morgado PJ, Suarez JA, Gomez LG, Morgado PJ Jr. Histoclinical basis for a new classification of hemorrhoidal disease. Dis Colon Rectum. 1988 Jun;31(6):474-80. doi: 10.1007/BF02552621. PMID 3378471
- [Background] Pigot F, Siproudhis L, Allaert FA. Risk factors associated with hemorrhoidal symptoms in specialized consultation. Gastroenterol Clin Biol. 2005 Dec;29(12):1270-4. doi: 10.1016/s0399-8320(05)82220-1. PMID 16518286
- [Background] Riss S, Weiser FA, Schwameis K, Riss T, Mittlbock M, Steiner G, Stift A. The prevalence of hemorrhoids in adults. Int J Colorectal Dis. 2012 Feb;27(2):215-20. doi: 10.1007/s00384-011-1316-3. Epub 2011 Sep 20. PMID 21932016
- [Background] Simillis C, Thoukididou SN, Slesser AA, Rasheed S, Tan E, Tekkis PP. Systematic review and network meta-analysis comparing clinical outcomes and effectiveness of surgical treatments for haemorrhoids. Br J Surg. 2015 Dec;102(13):1603-18. doi: 10.1002/bjs.9913. Epub 2015 Sep 30. PMID 26420725
- [Background] CRETON D. et le groupe closure®.Oblitération tronculaire saphène par le procédé radiofréquence VNUS Closure ®. résultats à 5 ans de l'étude multicentrique prospective,Phlébologie 2006,59 :67-72
- [Background] Becq A, Camus M, Rahmi G, de Parades V, Marteau P, Dray X. Emerging indications of endoscopic radiofrequency ablation. United European Gastroenterol J. 2015 Aug;3(4):313-24. doi: 10.1177/2050640615571159. PMID 26279839
- [Background] VIVALDI.C,. TOLKSDORFS. SCHAFER H., Radiofrequency ablation of hemorroïds. First results of a new technique The Rafaelo Procedure.Endarmpraxis;Colorectal disease 2017, 19 (suppl 2) p.138
- [Background] BORD C., PILLANT H., FAVREAU-WELTZER C., SENEJOUX A., SOUDAN D., ARREDONDO BISONO T., ZKIK A., BERDEAU G., ABRAMOWITZ L. Development of A Validated Questionnaire Evaluating The Burden of The Haemorrhoidal Disease and Anal Fissure (Hemo-Fiss). Value in Health, VOLUME 18, ISSUE 7, PA630, NOVEMBER 01, 2015